CLINICAL TRIAL: NCT04963036
Title: Impact of Nociception Level (NOL)-Guided Remifentanil Infusion and Entropy-guided Propofol Infusion on Intraoperative Arterial Pressure and Vasopressor Necessity A Prospective, Randomized, Controlled Trial.
Brief Title: Impact of Nociception Level (NOL)-Guided Remifentanil Infusion on Intraoperative Arterial Pressure and Vasopressor Necessity
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Centre Hospitalier Universitaire Saint Pierre (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: B0762021210506
Record Dates: First submitted 2021-06-14; First posted 2021-07-15 (Actual); Last update posted 2022-04-15 (Actual); Status verified 2021-07

CONDITIONS: Head and Neck Surgery; Maxillofacial Surgery
Keywords: Nociception; Entropy; Analgesia; Goal Directed Anesthesia Therapy (GDAT); Remifentanil; Intraoperative Hypotension; Myocardial Injury in Non-Cardiac Surgery (MINS); Postoperative Cognitive Dysfunction (POCD)
MeSH Terms: conditions — Agnosia; Postoperative Cognitive Complications | interventions — Entropy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Entropy and NOL-Guided Goal Directed Anesthesia (Experimental)
  Interventions: Other: Entropy and NOL-Guided Goal Directed Anesthesia
- Standard of Care Group (Entropy and blinded NOL) (Active Comparator)
  Interventions: Other: Standard of Care Group (Entropy and blinded NOL)

INTERVENTIONS:
Other: Entropy and NOL-Guided Goal Directed Anesthesia — Entropy-guided Anesthesia (Propofol infusion in order to maintain Entropy between 45 and 55) and NOL-guided Analgesia (Remifentanil infusion in order to maintain NOL-Index between 10 and 25).
  Arms: Entropy and NOL-Guided Goal Directed Anesthesia
Other: Standard of Care Group (Entropy and blinded NOL) — Entropy-guided Anesthesia (Propofol infusion in order to obtain Entropy between 45 and 55) and Remifentanil infusion at the discretion of the anesthetist in charge, based on current practice: patient vitals (Heart Rate, Blood Pressure, Respiratory Rate…), movements, spontaneous breathing, experience....
  In this group, nociception monitor screen will be concealed and the NOL index will not be available for guidance of remifentanil dosing).
  Arms: Standard of Care Group (Entropy and blinded NOL)

SUMMARY:
The aim of this study is to determine if Nociception Level (NOL)-guided Remifentanil analgesia, combined with Entropy-guided Propofol anesthesia, has a significant beneficial effect on the incidence of intraoperative hypotension episodes and/or on vasopressor requirements, during long-lasting major surgeries for high risk patients. The investigator will also investigate the effects of guided anesthesia on postoperative Myocardial Injury in Non-cardiac Surgery (MINS) and Postoperative cognitive dysfunction (POCD), amongst other frequent postoperative complications, in this population.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥18
* Elective high-risk head and neck or maxillo-facial surgery

Exclusion Criteria:

* Patient refusal
* Reduced ejection fraction below 40% and heart failure
* History of atrial Fibrillation, pulmonary embolism, recent cardioversion, recent cardiac ischemic episode, chronic hypotension, chronic kidney insufficiency (serum creatinine > 1.5)
* Septic state
* Baseline heart-rate < 50 or > 90 bpm
* History of psychiatric disease or medication

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2021-07-28 (Actual); Primary Completion 2022-06 (Estimated); Study Completion 2022-06 (Estimated)

PRIMARY OUTCOMES:
Occurrence of intraoperative hypotension | during surgery
  Occurrence of intraoperative hypotension is defined by at least 1 minute under the hypotension thresholds.
  Moderate and Severe Hypotension are respectively defined as a Mean Blood Pressure <65 mmHg or <55 mmHg and <75 or <65 mmHg for patient with history of chronic hypertension
Total Vasopressor Dose | during surgery
  Total Vasopressor Dose used throughout the intervention to maintain Arterial Pressure within a pre-defined individualized ranges (≥ 65 mmHg or ≥75 mmHg for patient with history of chronic hypertension, and ≤ 100 mmHg)
Number of interventions to cure intraoperative hypotension | during surgery
  Number of vasopressor boli or vasopressor infusion dose adjustments
Total Time under hypotension thresholds | during surgery
  Hypotension Thresholds ( <65 mmHg or < 75mmHg for patient with history of chronic hypertension)

SECONDARY OUTCOMES:
Myocardial Injury in Non-Cardiac Surgery (MINS) marker (Troponin T) | up to 48 hours after surgery
  Troponin T level measured before surgery, at end of surgery, 4 hours, 8 hours, 24 hours, 36 hours and 48 hours after surgery. The threshold is a postoperative concentration ≥ 20 ng/L with an increase from baseline of at least 5 ng/L, or a postoperative concentration ≥ 65 ng/L.
Postoperative Acute Kidney Injury (AKI) marker (creatinin/Glomerular Filtration Rate) | up to 48 hours after surgery
  Creatinin level measured before surgery, at end of surgery, 24 hours and 48 hours after surgery. The thresholds are defined by the Kidney Disease: Improving Global Outcomes (KDIGO) classification without the oliguria criteria.
Postoperative Cognitive Decline (POCD) | up to 6 months after surgery
  POCD will be evaluated by cognitive dysfunction battery tests (written Montreal Cognitive Assessment (MOCA) Test) at days 5,10, 15, hospital discharge, 3 and 6 postoperative months
PostOperative Delirium (PO Delirium) | up to 6 months after surgery
  PO Delirium will be evaluated by the Confusion Assessment Method (CAM) at days 5, 10, 15, hospital discharge, 3 and 6 postoperative months
Dosage of Stress Hormones | up to 4 hours after surgery
  Adrenocorticotropic Hormone (ACTH) and Cortisol will be measured in blood samples at the end of surgery, at the arrival in the ICU and at 4 hours after surgery.
Dosage of Neuro-Inflammatory Markers | up to 48 hours after surgery
  Interleukine-6 and Interleukine-8 will be measured in blood and saliva samples before surgery and during the postoperative period (4 hours, 24 hours and 48 hours after surgery).
Olfactory Function assessment as an indicator of Neuro-Inflammation | up to 48 hours after surgery
  A rapid quantitative olfactory function test, the University of Pennsylvania Smell Identification -Test (UPSIT-Test) will be performed before surgery and during the postoperative period (4 hours, 24 hours and 48 hours after surgery).
Length of Intensive Unit Care (IUC) stay | up to 10 Days after surgery
Length of hospital stay | up to 15 Days after surgery
Adverse Event (blood loss, infection) | up to 15 Days after surgery

CONTACTS AND LOCATIONS:
Overall Officials: Panayota Kapessidou, MD,PhD, Study Director — University Hospital Saint-Pierre (CHU Saint-Pierre), Université Libre de Bruxelles (ULB); Mehdi M'rini, MD, Principal Investigator — University Hospital Saint-Pierre (CHU Saint-Pierre), Université Libre de Bruxelles (ULB)
Locations (1):
- CHU Saint-Pierre, Brussels, Belgium

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Saugel B, Sessler DI. Perioperative Blood Pressure Management. Anesthesiology. 2021 Feb 1;134(2):250-261. doi: 10.1097/ALN.0000000000003610. No abstract available. PMID 33206118
- [Background] Sessler DI, Khanna AK. Perioperative myocardial injury and the contribution of hypotension. Intensive Care Med. 2018 Jun;44(6):811-822. doi: 10.1007/s00134-018-5224-7. Epub 2018 Jun 4. PMID 29868971
- [Background] Ruetzler K, Khanna AK, Sessler DI. Myocardial Injury After Noncardiac Surgery: Preoperative, Intraoperative, and Postoperative Aspects, Implications, and Directions. Anesth Analg. 2020 Jul;131(1):173-186. doi: 10.1213/ANE.0000000000004567. PMID 31880630
- [Background] Krzych LJ, Pluta MP, Putowski Z, Czok M. Investigating Association between Intraoperative Hypotension and Postoperative Neurocognitive Disorders in Non-Cardiac Surgery: A Comprehensive Review. J Clin Med. 2020 Sep 30;9(10):3183. doi: 10.3390/jcm9103183. PMID 33008109
- [Background] Feng X, Hu J, Hua F, Zhang J, Zhang L, Xu G. The correlation of intraoperative hypotension and postoperative cognitive impairment: a meta-analysis of randomized controlled trials. BMC Anesthesiol. 2020 Aug 5;20(1):193. doi: 10.1186/s12871-020-01097-5. PMID 32758153
- [Background] Greaves D, Psaltis PJ, Davis DHJ, Ross TJ, Ghezzi ES, Lampit A, Smith AE, Keage HAD. Risk Factors for Delirium and Cognitive Decline Following Coronary Artery Bypass Grafting Surgery: A Systematic Review and Meta-Analysis. J Am Heart Assoc. 2020 Nov 17;9(22):e017275. doi: 10.1161/JAHA.120.017275. Epub 2020 Nov 7. PMID 33164631
- [Background] Belrose JC, Noppens RR. Anesthesiology and cognitive impairment: a narrative review of current clinical literature. BMC Anesthesiol. 2019 Dec 27;19(1):241. doi: 10.1186/s12871-019-0903-7. PMID 31881996
- [Background] Walsh M, Devereaux PJ, Garg AX, Kurz A, Turan A, Rodseth RN, Cywinski J, Thabane L, Sessler DI. Relationship between intraoperative mean arterial pressure and clinical outcomes after noncardiac surgery: toward an empirical definition of hypotension. Anesthesiology. 2013 Sep;119(3):507-15. doi: 10.1097/ALN.0b013e3182a10e26. PMID 23835589
- [Background] Evered LA, Silbert BS. Postoperative Cognitive Dysfunction and Noncardiac Surgery. Anesth Analg. 2018 Aug;127(2):496-505. doi: 10.1213/ANE.0000000000003514. PMID 29889707
- [Background] Ledowski T. Monitoring nociception-getting 'there yet' might be easier with a road map. Br J Anaesth. 2017 Oct 1;119(4):716-717. doi: 10.1093/bja/aex277. No abstract available. PMID 29121306
- [Background] Ledowski T. Objective monitoring of nociception: a review of current commercial solutions. Br J Anaesth. 2019 Aug;123(2):e312-e321. doi: 10.1016/j.bja.2019.03.024. Epub 2019 Apr 30. PMID 31047645
- [Background] De Jonckheere J, Bonhomme V, Jeanne M, Boselli E, Gruenewald M, Logier R, Richebe P. Physiological Signal Processing for Individualized Anti-nociception Management During General Anesthesia: a Review. Yearb Med Inform. 2015 Aug 13;10(1):95-101. doi: 10.15265/IY-2015-004. PMID 26293855
- [Background] Martini CH, Boon M, Broens SJ, Hekkelman EF, Oudhoff LA, Buddeke AW, Dahan A. Ability of the nociception level, a multiparameter composite of autonomic signals, to detect noxious stimuli during propofol-remifentanil anesthesia. Anesthesiology. 2015 Sep;123(3):524-34. doi: 10.1097/ALN.0000000000000757. PMID 26154185
- [Background] Meijer F, Honing M, Roor T, Toet S, Calis P, Olofsen E, Martini C, van Velzen M, Aarts L, Niesters M, Boon M, Dahan A. Reduced postoperative pain using Nociception Level-guided fentanyl dosing during sevoflurane anaesthesia: a randomised controlled trial. Br J Anaesth. 2020 Dec;125(6):1070-1078. doi: 10.1016/j.bja.2020.07.057. Epub 2020 Sep 17. PMID 32950246
- [Background] Futier E, Lefrant JY, Guinot PG, Godet T, Lorne E, Cuvillon P, Bertran S, Leone M, Pastene B, Piriou V, Molliex S, Albanese J, Julia JM, Tavernier B, Imhoff E, Bazin JE, Constantin JM, Pereira B, Jaber S; INPRESS Study Group. Effect of Individualized vs Standard Blood Pressure Management Strategies on Postoperative Organ Dysfunction Among High-Risk Patients Undergoing Major Surgery: A Randomized Clinical Trial. JAMA. 2017 Oct 10;318(14):1346-1357. doi: 10.1001/jama.2017.14172. PMID 28973220
- [Background] Meijer FS, Martini CH, Broens S, Boon M, Niesters M, Aarts L, Olofsen E, van Velzen M, Dahan A. Nociception-guided versus Standard Care during Remifentanil-Propofol Anesthesia: A Randomized Controlled Trial. Anesthesiology. 2019 May;130(5):745-755. doi: 10.1097/ALN.0000000000002634. PMID 30829658
- [Background] Salmasi V, Maheshwari K, Yang D, Mascha EJ, Singh A, Sessler DI, Kurz A. Relationship between Intraoperative Hypotension, Defined by Either Reduction from Baseline or Absolute Thresholds, and Acute Kidney and Myocardial Injury after Noncardiac Surgery: A Retrospective Cohort Analysis. Anesthesiology. 2017 Jan;126(1):47-65. doi: 10.1097/ALN.0000000000001432. PMID 27792044
- [Background] Sessler DI, Bloomstone JA, Aronson S, Berry C, Gan TJ, Kellum JA, Plumb J, Mythen MG, Grocott MPW, Edwards MR, Miller TE; Perioperative Quality Initiative-3 workgroup; POQI chairs; Miller TE, Mythen MG, Grocott MP, Edwards MR; Physiology group; Preoperative blood pressure group; Intraoperative blood pressure group; Postoperative blood pressure group. Perioperative Quality Initiative consensus statement on intraoperative blood pressure, risk and outcomes for elective surgery. Br J Anaesth. 2019 May;122(5):563-574. doi: 10.1016/j.bja.2019.01.013. Epub 2019 Feb 27. PMID 30916004
- [Background] Danielson M, Wiklund A, Granath F, Blennow K, Mkrtchian S, Nellgard B, Oras J, Jonsson Fagerlund M, Granstrom A, Schening A, Rasmussen LS, Erlandsson Harris H, Zetterberg H, Ricksten SE, Eriksson LI. Neuroinflammatory markers associate with cognitive decline after major surgery: Findings of an explorative study. Ann Neurol. 2020 Mar;87(3):370-382. doi: 10.1002/ana.25678. Epub 2020 Jan 25. PMID 31930549